CLINICAL TRIAL: NCT03346187
Title: A Randomized, Open-label, Single Oral Dose, 2-way Crossover Clinical Trial to Compare Safety and Pharmacokinetic Characteristics of CKD-337 in Healthy Male Volunteers
Brief Title: A Clinical Trial to Compare Safety and Pharmacokinetic Characteristics of CKD-337
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 146BE16007
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Period 1: Active Comparator(Atorvastatin Calcium Trihydrate+Fenofibrate), 2 tablets administered under fed conditions.
  Period 2: test drug(CKD-337 : Atorvastatin Calcium Trihydrate + Fenofibrate), 1 capsule administered under fed conditions.
  Interventions: Drug: Active Comparator(Atorvastatin Calcium Trihydrate+Fenofibrate); Drug: Test drug(CKD-337)
- B (Experimental): Period 1: test drug(CKD-337 : Atorvastatin Calcium Trihydrate + Fenofibrate), 1 capsule administered under fed conditions.
  Period 2: Active Comparator(Atorvastatin Calcium Trihydrate+Fenofibrate), 2 tablets administered under fed conditions.
  Interventions: Drug: Active Comparator(Atorvastatin Calcium Trihydrate+Fenofibrate); Drug: Test drug(CKD-337)

INTERVENTIONS:
Drug: Active Comparator(Atorvastatin Calcium Trihydrate+Fenofibrate) — Lipitor(Atorvastatin Calcium Trihydrate 20mg/tablet) + Lipidil supra(Fenofibrate 160mg/tablet)
Drug: Test drug(CKD-337) — CKD-337(Atorvastatin calcium trihydrate 20mg+choline fenofibrate 178.8mg/capsule)

SUMMARY:
A randomized, open-label, single oral dose, 2-way crossover clinical trial to compare safety and pharmacokinetic characteristics of CKD-337 in healthy male volunteers

DETAILED DESCRIPTION:
This study is a randomized, open-label, single oral dose, 2-way crossover clinical trial to compare safety and pharmacokinetics of CKD-337 in healthy male volunteers.

Subjects will receive either a single oral dose of the test formulation(CKD-337) or a oral dose of the reference formulation(Atorvastatin Calcium Trihydrate+Fenofibrate).

Each treatment period was separated by a washout period of at least 7 days.

ELIGIBILITY:
* Inclusion Criteria:

  1. Healthy male older than 19 years and under 45 years at the time of screening
  2. BMI 17.5~30.5 kg/m² and body weight more than 55kg

     * BMI = Weight(kg)/{Height(m)}²
  3. Subject who is no chronic disease, no symptoms or pathological findings
  4. Suitable subject who is determined by laboratory tests(hematology test, blood chemistry, urinalysis test etc.), Vital Sign, ECG test at the time of screening
  5. Subject who fully understand the clinical trials after in-depth explanation, decide to join the clinical trials and sign on an inform consent from willing
* Exclusion Criteria:

  1. Subject who has a clinically significant disease such as hepatic, kidneys, neurological, respiratory, endocrine, hemato-oncology, urinary, cardiovascular, musculoskeletal or psychiatric diseases and who has a following history

     * Gallbladder disease including cholelithiasis, severe hepatic impairment
     * Acute/chronic pancreatitis due to hypertriglyceridemia
     * Pulmonary embolism or interstitial lung disease
     * Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
     * Hypoalbuminemia
     * Alcoholics
     * Predisposition to rhabdomyolysis
  2. Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect drug absorption
  3. Subject who has hypersensitivity to the drug composition containing choline fenofibrate, fenofibrate or atorvastatin, and other drug(aspirin, fenofibrate series, antibiotic and so on)
  4. The following clinical significant findings in the EKG at the time of screening

     * QTc(Q-T interval corrected for heart rate) > 450ms
     * PR interval(The interval between the beginning of the P wave and the beginning of the QRS complex in ECG) > 200msec
     * QRS duration(The duration of the Q,R and S wave in ECG) > 120msec
  5. The following results in the clinical laboratory tests

     * CPK(Creatinine Phospho-Kinase) > 2 x upper limit of normal range
     * Liver function test(AST; Aspartate Transaminase, ALT; Alanine Transaminase, ALP; Alkaline phosphatase, Total bilirubin, γ-GT) > 2 x upper limit of normal range
     * eGFR(Estimated Glomerular Filtration Rate) < 60 mL/min/1.73m² Calculated by MDRD(Modification of Diet in Renal Disease)
  6. Systolic blood pressure ≥ 160mmHg(millimeter of mercury) or ≤ 100mmHg(millimeter of mercury) , Diastolic blood pressure ≥ 95mmHg(millimeter of mercury) or ≤ 60mmHg(millimeter of mercury) at the time of screening
  7. History of drug abuse or a positive reaction for drug abuse in the urine at the time of screening
  8. Taking medicines that are known to significantly induce or inhibit drug metabolizing enzymes, including barbiturates, within 30 days of the first dosing
  9. Those who experience photoallergy or phototoxicity during treatment with fibrates or ketoprofen
  10. Taking ETC(Ethical Drug), oriental medicine within 2 weeks and OTC(Over-the-counter Drug), vitamin within 10 days before the first dosing
  11. Taking the medication involved in other clinical trials within 3 months before the first dosing
  12. Whole blood donation with 2 months, component blood donation or blood transfusion within 1 month before the first dosing
  13. Alcohol > 21 units/week (1unit=10g of pure alcohol), continuously within 6 month before the first dosing or Who can not stop drinking alcohol during the clinical trial
  14. Smoker(> 10 cigarettes/day) for the last 3 months or who can not stop smoking during the clinical trial
  15. Consumption of food containing grapefruit within 48 hours before first dosing and who can not stop consumption it until EOS(End of study)
  16. Consumption of food containing caffeine(e.g. coffee, green tea etc.) within 24 hours before first dosing and who can not stop consumption it until discharge
  17. Not using a reliable contraception or planning a pregnancy during the clinical trial
  18. Unsuitable Conditions including laboratory result by investigator's judgement

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Atorvastatin AUCt(Area under the plasma drug concentration-time curve) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration]
Atorvastatin Cmax(Maximum plasma concentration) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Fenofibric acid AUCt | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Cmax | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration

SECONDARY OUTCOMES:
Atorvastatin AUCinf(Area under plasma concentration-time curve from time point of administration to infinite) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin Tmax(Time taken to reach the maximum concentration) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin t1/2(Terminal half-life, Time for Cmax to drop in half) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin CL/F(Apparent total body clearance after extravascular administration, calculated as Dose/AUC) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Atorvastatin Vd/F(Apparent volume of distribution/Bioavailability) | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
Fenofibric acid AUCinf | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Tmax | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid t1/2 | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid CL/F | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
Fenofibric acid Vd/F | Predose(0hr), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96hr after drug administration
2-hydroxy atorvastatin AUCt | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Cmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin AUCinf | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Tmax | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin t1/2 | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin CL/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration
2-hydroxy atorvastatin Vd/F | Predose(0hr), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48hr after drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University Hospital, Busan, Seo-gu, South Korea